CLINICAL TRIAL: NCT04598516
Title: Maastricht Investigation of Renal Function in Absence of- and Post- Contrast in Patients With Estimated Glomerular Filtration Rate LEss Than 30mL/Min/1.73m2
Brief Title: Maastricht Investigation of Renal Function in Absence of- and Post- Contrast in Patients With eGFR LEss Than 30
Acronym: MIRACLE
Status: Withdrawn | Type: Observational
Why Stopped: delay
Sponsor: Maastricht University Medical Center (Other)
Responsible Party: Sponsor
Other Study IDs: NL.MUMC.AMACINGrp.1
Record Dates: First submitted 2020-10-07; First posted 2020-10-22 (Actual); Last update posted 2023-10-19 (Actual); Status verified 2023-10

CONDITIONS: Acute Kidney Injury (Nontraumatic); Contrast-induced Nephropathy; Renal Insufficiency
Keywords: intravascular iodinated contrast; Post-Contrast Acute Kidney Injury; Contrast-induced acute kidney injury
MeSH Terms: conditions — Acute Kidney Injury; Renal Insufficiency

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — serum samples may be stored for renal damage biomarker assays
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: serum creatinine assay — peak change in serum creatinine in a period of 5 days from baseline (day 0) will be determined

SUMMARY:
Intravascular iodinated contrast administration has become crucial to modern medicine. Currently it is estimated that over 250 million injections are given each year worldwide during medical scans and interventions. An acute predefined increase in serum creatinine is considered an indicator of acute kidney injury (AKI). When such an acute increase in serum creatinine occurs within 5 days post-contrast in absence of another aetiology, it is assumed to be iodinated contrast administration induced acute kidney injury. For over 50 years now, acute kidney injury caused by intravascular administration of iodinated contrast material has been considered a leading cause of hospital-acquired renal failure. Contrast has been withheld in fear of kidney injury with misdiagnoses and delayed appropriate patient management as a result. Since 2018, it is now widely accepted that only patients with eGFR <30 mL/min/1.73m2 are at risk of renal injury after intravascular iodinated contrast material injection. However, no study to date has been able to distinguish acute kidney injury caused by iodinated contrast administration from that for which no causal link is established, and it is unsure a causal relationship exists. There are several studies, in attempts to evaluate the causal relationship between contrast exposure and nephrotoxicity, that found fluctuations in absence of contrast similar to those considered to be contrast-induced acute kidney injury. Similarly, it is unsure whether longer-term negative outcomes are inherent to the population studied or a result of contrast administration. However, most of these studies are observational and retrospective in nature. The issue with retrospective studies is that they often cannot control for confounders and therefore cannot give us causation, only association. On the other hand, prospective randomized controlled trials comparing intravascular iodinated contrast administration to no contrast are unlikely given evident ethical issues. The current prospective observational study proposes to use intra-patient comparisons of peak change in renal function during periods in absence of- and with contrast to elucidate the relationship between renal function and contrast administration in this population.

DETAILED DESCRIPTION:
The current prospective observational study proposes to use intra-patient comparisons of peak changes in renal function (serum creatinine) in absence of- and post- intravascular iodinated contrast administration, to elucidate the relationship between renal function and contrast administration in elective patients with eGFR <30 mL/min/1.73m2. The effects of contrast administration on risk of 1-month dialysis and mortality will also be evaluated.

Daily serum creatinine assays will be done 1. during 5 days before contrast (= in absence of contrast), 2. during 5 days after contrast (= post-contrast), and 3. during 5 days at 1-month post contrast (= 1-month post contrast in absence of contrast). Baseline serum creatinine values will be obtained on the day before each 5-day series.

Relevant baseline characteristics of patients will be reported to enable a detailed description of the study population. To explore whether the magnitude of the mean difference in peak change in serum creatinine before and after contrast administration depends on other factors, pre-planned subgroup analyses will be performed. To enable subgroup analyses, data will be collected on 1) prophylactic hydration (yes vs no); 2) administration route (intra-arterial versus intravenous contrast administration); 3) contrast volume (high vs low) and 4) comorbidity (presence vs absence of diabetes).

ELIGIBILITY:
Inclusion Criteria:

* eGFR <30 mL/min/1.73m2 in absence of dialysis
* referred for an elective procedure with intravascular administration of iodinated contrast material at Maastricht UMC+

Exclusion Criteria:

* age <18 years
* dialysis or pre-dialysis
* intravascular contrast administration <30 days before the first baseline measurement
* emergency or intensive care status
* inability to complete follow-up

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with eGFR <30 mL/min/1.73m2 in absence of dialysis referred for an elective procedure with intravascular administration of iodinated contrast material at Maastricht UMC+ are eligible for inclusion.
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2097-11-01 (Estimated); Primary Completion 2099-11-01 (Estimated); Study Completion 2099-11-01 (Estimated)

PRIMARY OUTCOMES:
Mean difference in peak change in serum creatinine from baseline between a 5 day period before contrast and a 5 day period immediately after contrast. | 5 days
  The underlying hypothesis is that intravascular iodinated contrast administration will cause greater peak changes in serum creatinine within 5 days. The primary outcome is peak changes in serum creatinine within 5 days from a baseline measurement. The effect of contrast administration will be expressed as the mean intra-patient difference in peak changes in serum creatinine between pre- and post-contrast periods. Peak change in eGFR will also be calculated based on the peak serum creatinine values.

SECONDARY OUTCOMES:
Mean difference in peak change in serum creatinine from baseline between a 5 day period before contrast and a 5 day period at 1-month post-contrast. | 5 days
  mean intra-patient difference between peak changes in serum creatinine occurring within 5 days pre-contrast and 5 days at 1-month post-contrast from baseline measurements (baseline = measurement on the day before every 5-day series). Peak change in eGFR will also be calculated based on the peak serum creatinine values.
Time to post-contrast peak change in serum creatinine. | 5 days
  Time to greatest post-contrast change in serum creatinine from baseline (day 0) within 5 days after contrast administration.
Acute kidney injury in absence of- vs post-contrast. | 5 days
  Incidences of peak changes in serum creatinine corresponding to definitions for classic CIN (an increase in serum creatinine greater than 44umol/l or greater than 25% from baseline) and KDIGO acute kidney injury (an increase in serum creatinine greater than 26.5 umol/L from baseline or more than 1.5 times the baseline value). Peak changes will be determined within 5 days pre-contrast and 5 days post-contrast.
1 month eGFR decline >=5 mL/min/1.73m2. | 1 month, 1 year
  Incidences of peak eGFR decline >=5 mL/min/1.73m2 within 5 days pre- and within 5 days at 1-month post-contrast
1 month dialysis and mortality. | 1 month
  Incidences of dialysis and mortality at 1 month post-contrast.

CONTACTS AND LOCATIONS:
Locations (1):
- Maastricht UMC, Maastricht, Netherlands

IPD SHARING:
Plan to Share IPD: No